CLINICAL TRIAL: NCT01637987
Title: Nurse Peripheral Intravenous Catheter Insertion Success With and Without Assistive Devices in Patients 0-12 Months of Age
Brief Title: Nurse PIV Insertion Success With and Without Assistive Devices in Patients 0-12 Months of Age
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Combination of insufficient research staff support, insufficient subjects meeting enrollment criteria, and investigators changing role responsibilities. Administratively closed (continuing review or completion report not submitted).
Sponsor: University of Nebraska (Other)
Collaborators: Children's Hospital and Medical Center, Omaha, Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0694-11-EP
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: PIV Catheter Insertion; Vein Visualization
Keywords: Peripheral intravenous catheter; Vein visualization; Transillumination; Near infrared light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unassisted vein visualization (Active Comparator): The traditional technique of vein visualization and palpation will be used to identify veins during peripheral intravenous line (PIV) insertion procedures. This involves the use of a tourniquet to facilitate venous pooling to see the vein and prevent vein rupture during cannulation. Nurse may use heat application to facilitate vein identification.
  Interventions: Procedure: Unassisted vein visualization
- Wee Sight Transilluminator (Active Comparator): The Wee Sight® Transilluminator (Philips Children's Medical Ventures, Monroeville, PA) is a hand held, non-heat producing, light emitting diode (Class 2), battery operated device. The device assists in vein identification by being held adjacent to or under the subject's extremity to visualize the venous anatomy superficial veins absorb light and appear as dark lines against the surrounding illuminated tissues. This will be used to identify veins during peripheral intravenous line (PIV) insertion procedures.
  Interventions: Procedure: Wee Sight® Transilluminator
- Near Infra-red light (VeinViewer) (Active Comparator): VeinViewer near infrared light views hemoglobin up to 10 mm beneath skin. Hemoglobin absorbs the light while surrounding tissue scatters it providing a suitable contrast between the vein & surrounding subcutaneous tissue. This data is captured, digitally processed by video camera, and projected back onto the skin as a visual image of venous anatomy. This will be used to identify veins during peripheral intravenous line (PIV) insertion procedures.
  Interventions: Procedure: VeinViewer® (Christie Digital Systems, Cypress, CA)

INTERVENTIONS:
Procedure: Unassisted vein visualization — The traditional technique of vein visualization and palpation will be used to identify veins during the PIV insertion procedures. This involves the use of a tourniquet to facilitate venous pooling to see the vein and prevent vein rupture during cannulation. Nurse may use heat application to facilitate vein identification.
  Other Names: Traditional methods of vein identification
  Arms: Unassisted vein visualization
Procedure: Wee Sight® Transilluminator — The Wee Sight® Transilluminator (Philips Children's Medical Ventures, Monroeville, PA) is a hand held, non-heat producing, light emitting diode (Class 2), battery operated device. The device is held adjacent to or under the subject's extremity to visualize the venous anatomy superficial veins absorb light and appear as dark lines against the surrounding illuminated tissues. Vein visualization improves with dimmed room lighting and a thin subcutaneous tissue layer. Nurse will assess vascular anatomy using traditional techniques of visualization and palpation with tourniquet/heat application as needed, and add the Wee Sight to assist in vein identification.
  Other Names: Vein Transillumination
  Arms: Wee Sight Transilluminator
Procedure: VeinViewer® (Christie Digital Systems, Cypress, CA) — VeinViewer near infrared light views hemoglobin up to 10 mm beneath skin. Hemoglobin absorbs the light while surrounding tissue scatters it providing a suitable contrast between the vein & surrounding subcutaneous tissue. This data is captured, digitally processed by video camera, and projected back onto the skin as a visual image of venous anatomy. Nurse will assess vascular anatomy using traditional techniques of visualization and palpation with tourniquet/heat application as needed, and add the VeinViewer to assist in vein identification.
  Other Names: Vein Viewer
  Arms: Near Infra-red light (VeinViewer)

SUMMARY:
The purpose of this study is to determine if the use of a vein identification assistive device increases nurse PIV insertion success within the first two attempts in children 0-12 months of age when compared to unassisted methods.

DETAILED DESCRIPTION:
Obtaining peripheral intravenous (PIV) access is a nearly universal procedure for medical management of the hospitalized pediatric patient. In children, PIV placement can often be difficult due to the inability to identify peripheral veins (Wilson, 2007). Many assistive devices have been used or promoted to improve vein visualization with the intention of increasing PIV insertion success. Limited research was found to support this assumption regarding nursing PIV insertion success in children. This study is a randomized, controlled trial to determine if the use of a vein identification assistive device increases nurse PIV insertion success within the first two attempts in children 0-12 months of age when compared to unassisted methods. Patients admitted to Children's Hospital & Medical Center (CHMC) Emergency Department, 4th floor medical-surgical unit, or 5th floor medical-surgical/ Intermediate Care Unit, up to 12 months of age requiring non-emergent PIV placement as part of their medical plan of care will be eligible. Following consent subjects will be randomized into one of three vein identification method study groups (1) Wee Sight Transilluminator - a hand held light emitting device held adjacent to or under the patient's extremity to visualize the venous anatomy; (2) VeinViewer - uses near infrared light to view hemoglobin and projects an image of venous anatomy onto the skin; and (3) Unassisted Methods - traditional techniques of vein visualization and palpation. Based on study group assignment the nurse will use the appropriate vein identification method during the first two PIV insertion attempts. Evaluation of vein identification methods will be based on PIV insertion success or failure.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Children's Hospital & Medical Center Emergency Department, 4th floor medical-surgical unit, or 5th floor medical-surgical/Intermediate Care Unit
* Require non-emergent PIV placement as part of medical plan of care
* Less than or equal to 12 month birth date

Exclusion Criteria:

* Greater than 12 month birth date
* PIV not required
* PIV inserted by practitioner other than RN
* PIV inserted by RN not employed by study areas
* Ward of state
* Require emergent PIV placement
* Primary language is not English or Spanish

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Successful PIV insertion during first or second cannulation attempt. | Immediate upon completing first or second PIV insertion attempt
  Success = Insertion of a 22 or 24-gauge catheter into a peripheral vein followed by the immediate ability to flush 1-2 ml normal saline without signs of venous infiltration (e.g., pain and swelling).
  Failure = Inability to insert a 22 or 24-gauge catheter into a peripheral vein, or insertion of a catheter into a peripheral vein followed by the immediate inability to flush 1-2 ml normal saline or signs of infiltration upon flushing.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Peterson, MSN, Principal Investigator — Children's Hospital and Medical Center, Omaha, NE
Locations (1):
- Children's Hospital and Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Peterson KA, Phillips AL, Truemper E, Agrawal S. Does the use of an assistive device by nurses impact peripheral intravenous catheter insertion success in children? J Pediatr Nurs. 2012 Apr;27(2):134-43. doi: 10.1016/j.pedn.2010.10.009. Epub 2011 Feb 18. PMID 22341192
- [Background] Chapman LL, Sullivan B, Pacheco AL, Draleau CP, Becker BM. VeinViewer-assisted Intravenous catheter placement in a pediatric emergency department. Acad Emerg Med. 2011 Sep;18(9):966-71. doi: 10.1111/j.1553-2712.2011.01155.x. Epub 2011 Aug 19. PMID 21854488
- [Background] Perry AM, Caviness AC, Hsu DC. Efficacy of a near-infrared light device in pediatric intravenous cannulation: a randomized controlled trial. Pediatr Emerg Care. 2011 Jan;27(1):5-10. doi: 10.1097/PEC.0b013e3182037caf. PMID 21178814
- [Background] Hess HA. A biomedical device to improve pediatric vascular access success. Pediatr Nurs. 2010 Sep-Oct;36(5):259-63. PMID 21067078